CLINICAL TRIAL: NCT00484627
Title: Ergogenic Effects of Creatine Supplementation in HIV Infection
Brief Title: Effects of Creatine and Resistance Exercise Training in People With HIV Infection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: R01AT000491-01 (NIH)
Record Dates: First submitted 2007-06-08; First posted 2007-06-11 (Estimated); Last update posted 2007-06-11 (Estimated); Status verified 2007-06

CONDITIONS: HIV Infections
Keywords: Exercise; HIV; Creatine; Muscle
MeSH Terms: conditions — HIV Infections; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Use of creatine monohydrate (a dietary supplement)
Behavioral: Progressive resistance exercise training

SUMMARY:
This study was designed determine whether use of creatine monohydrate, a dietary supplement, can increase skeletal muscle mass and strength and improve the response to progressive resistance exercise training in people with HIV infection.

DETAILED DESCRIPTION:
This is a randomized, placebo-controlled study to evaluate the effect of creatine monohydrate, a dietary supplement, on skeletal muscle size and function (i.e., strength, energy metabolism, work capacity, fatigue); whole-body exercise performance; and body composition. This study is also designed to determine whether creatine supplementation augments the functional benefit derived from progressive resistance exercise. The safety of creatine supplementation in people with HIV infection will also be evaluated. Forty HIV-positive subjects will be randomly assigned, on a 1:1 basis, to receive creatine monohydrate or placebo for a period of 14 days, followed by a 12-week program of supervised progressive resistance exercise training during which administration of creatine monohydrate or placebo will continue.

Measurements of muscle strength, size, composition, energetics and fatigue, as well as body weight and composition and serum biochemistries, will be made at baseline, after two weeks of treatment with creatine or placebo (before PRT), and again after 12 weeks of PRT (study week 14). Safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Clinically stable, sedentary HIV-positive adults who are on optimized antiretroviral regimens and plan to remain so during the study.
* Men and women on hormone replacement therapy and women using hormonal contraceptives must have been on stable regimens for the preceding 6 months and plan to continue on such treatment throughout the study period.

Exclusion Criteria:

* Serum creatinine > 1.5 mg/dl or clinical evidence of renal disease or prior kidney transplant
* Creatine kinase (CK) > 1.5 times the upper limit of normal (ULN)
* Hemoglobin < 8.5 g/dl
* AST, ALT, or LDH > 5 X ULN
* Uncontrolled diarrhea (> 6 stools per day)
* Impaired oral intake
* Persistent nausea or vomiting
* Untreated hypogonadism
* Pharmacologic use of growth hormone, testosterone, oxandrolone, nandrolone decanoate, oxymetholone, or other oral, injectable, or transdermal anabolic steroids, androstenedione, or dehydroepiandrosterone (DHEA) within the preceding 6 months (subjects with documented hypogonadism on stable testosterone replacement, defined as a dose < 300 mg q2 weeks for the preceding 6 months, will be allowed to enroll)
* Use of glucocorticoids, megestrol acetate, creatine monohydrate, cytokine inhibitors (thalidomide, pentoxifylline, ketotifen), drugs known to adversely affect renal function, cytokines, parenteral or tube feeding, or initiation of treatment for a systemic infection within 30 days prior to enrollment
* History of angina, coronary heart disease, or congestive heart failure
* Current pregnancy or lactation or plans to become pregnant.
* Because vegetarians are known to have lower intramuscular concentrations of creatine and therefore may experience a much greater relative increase in muscle creatine levels, we will exclude such individuals from this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2001-08; Study Completion 2003-10 (Actual)

PRIMARY OUTCOMES:
Muscle strength | 14 weeks

SECONDARY OUTCOMES:
Muscle size | 14 weeks
Muscle energetics | 14 weeks
Body composition | 14 weeks
Biochemistries | 14 weeks
Safety | Throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: Morris Schambelan, MD, Principal Investigator — University of California, San Francisco; San Francisco General Hospital; Kathleen Mulligan, PhD, Study Director — University of California, San Francisco; San Francisco General Hospital
Locations (1):
- San Francisco General Hospital, San Francisco, California, United States

REFERENCES:
- [Derived] Sakkas GK, Mulligan K, Dasilva M, Doyle JW, Khatami H, Schleich T, Kent-Braun JA, Schambelan M. Creatine fails to augment the benefits from resistance training in patients with HIV infection: a randomized, double-blind, placebo-controlled study. PLoS One. 2009;4(2):e4605. doi: 10.1371/journal.pone.0004605. Epub 2009 Feb 26. PMID 19242554